CLINICAL TRIAL: NCT03585231
Title: Say "Hello" To Your Digital Coach: Development and Pilot Trial of the First Conversational Agent for Smoking Cessation
Brief Title: Pilot Trial of the First Conversational Agent for Smoking Cessation (QuitBot)
Acronym: QuitBot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8659; NCI-2018-03684 (Registry Identifier: NCI / CTRP); RG1001766 (Other: Fred Hutch/University of Washington Cancer Consortium); 8659 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2018-06-29; First posted 2018-07-12 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Smoking Cessation
Keywords: Smoking; Chatbot; Conversational agent; Chatbot for quitting smoking; Messaging; Text messaging; SMS
MeSH Terms: conditions — Smoking Cessation; Smoking

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental (Experimental): This is the experimental arm of the study. This includes receiving immediate access to the novel/experimental smoking cessation messaging program. Therapy description withheld to protect the integrity of the study.
  Interventions: Behavioral: Immediate access to novel messaging program intervention
- Control (Active Comparator): This is the control arm of the study. This includes receiving receiving immediate access to the standard of care smoking cessation messaging program. Therapy description withheld to protect the integrity of the study.
  Interventions: Behavioral: Immediate access to standard of care messaging program intervention
- Delayed Control (Active Comparator): This is the second control arm of the study. This includes receiving the novel/experimental smoking cessation messaging program after completing the 3-month follow-up survey. Therapy description withheld to protect the integrity of the study.
  Interventions: Behavioral: Delayed access to novel novel messaging program intervention

INTERVENTIONS:
Behavioral: Immediate access to novel messaging program intervention — The experimental arm includes an immediate intervention using a novel messaging program for smoking cessation.
  Arms: Experimental
Behavioral: Immediate access to standard of care messaging program intervention — The immediate control intervention uses a standard of care messaging program for smoking cessation.
  Arms: Control
Behavioral: Delayed access to novel novel messaging program intervention — The delayed control intervention uses the novel messaging program for smoking cessation.
  Arms: Delayed Control

SUMMARY:
Conversational agents (CAs) are computer-powered digital coaches designed to form long-term social-emotional connections with users through conversations. We have developed a CA for cigarette smoking cessation. In a pilot randomized trial (N = 415), we will compare the experimental messaging program (n = 155) with the standard of care national government smoking cessation messaging program (n = 157), and then we will compare immediate (n=51) versus delayed (n=51) access to the the experimental messaging program, to assess 12-week usability, receptivity, and preliminary cessation results in adults in western Washington State and nationally across the US who want to quit smoking.

DETAILED DESCRIPTION:
Cigarette smoking is the most preventable cause of cancer in the US, accounting for one-third of all cancer deaths. Within the Fred Hutchinson Center's western Washington State 13-county catchment area, there are enormous disparities in adult cigarette smoking rates. Our recently completed WebQuit website RCT for smoking cessation had low engagement and no personalization to users' needs. Fortunately, a potentially game-changing solution to the problems of engagement and lack of personalization provide a new direction for my research. Advances in machine learning, natural language processing, and cloud computing are making it possible to create and widely disseminate conversational agents (CAs), which are computer-powered digital coaches designed to form long-term social-emotional connections with users through conversations. We have developed a CA for cigarette smoking cessation. In a pilot randomized trial (N = 415), we will compare the experimental messaging program with the standard of care national government smoking cessation messaging program, and then we will compare immediate versus delayed access to the the experimental messaging program. Twelve-week usability, receptivity, and preliminary cessation results will provide critical and timely pilot data.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older
* smokes at least five cigarettes daily for at least past 12 months
* wants to quit cigarette smoking in the next 14 days
* if concurrently using any other nicotine or tobacco products, wants to quit using them within the next 14days
* resides in western Washington State (in the following counties: Clallam, Grays Harbor, Island, Jefferson, King, Kitsap, Mason, Pierce, San Juan, Skagit, Snohomish, Thurston, and Whatcom)
* interested in learning skills to quit smoking
* willing to be randomly assigned to either condition
* has at least daily access to their own personal smartphone
* has and uses both text messaging and Facebook Messenger on their smartphone
* willing and able to read in English
* not using other smoking cessation interventions (including apps or our other intervention studies).
* willing to complete one 3-month follow-up survey
* willing to provide email, phone, and mailing address.

Exclusion Criteria:

* The exclusion criteria are opposite of the inclusion criteria listed above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 404 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2019-12-06 (Actual); Study Completion 2020-12-02 (Actual)

PRIMARY OUTCOMES:
30-day point prevalence abstinence | 3 months post randomization
  No smoking in the past 30 days, as reported 3 month post treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Bricker, PhD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bricker JB, Sullivan B, Mull K, Santiago-Torres M, Lavista Ferres JM. Conversational Chatbot for Cigarette Smoking Cessation: Results From the 11-Step User-Centered Design Development Process and Randomized Controlled Trial. JMIR Mhealth Uhealth. 2024 Jul 23;12:e57318. doi: 10.2196/57318. PMID 38913882